CLINICAL TRIAL: NCT00136552
Title: FL-2000 Study for Newly Diagnosed Follicular Lymphoma Patients With a High Tumor Burden
Brief Title: Study for Newly Diagnosed Follicular Lymphoma Patients With a Large Tumor Burden
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Lymphoma Study Association (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: FL2000; PHRC
Record Dates: First submitted 2005-08-25; First posted 2005-08-29 (Estimated); Last update posted 2007-07-03 (Estimated); Status verified 2007-07

CONDITIONS: Lymphoma
Keywords: lymphoma; follicular; B-cell; rituximab; interferon
MeSH Terms: conditions — Lymphoma | interventions — Rituximab

INTERVENTIONS:
Drug: rituximab

SUMMARY:
The purpose of this study is to assess in a prospective multicentric study (Phase III) the introduction of a monoclonal antibody directed against B-cells associated with a standard therapy including chemotherapy and alpha-interferon in first line treatment of patients with a large tumor burden follicular lymphoma.

DETAILED DESCRIPTION:
Follicular lymphoma patients with a large tumor burden will be randomized for 18 months of treatment with either:

* Arm A: CHVP + alpha2a-interferon. Patients will receive 12 courses of CHVP (cyclophosphamide 600 mg/m², adriamycin 25 mg/m², etoposide 100 mg/m² on day 1 and prednisolone 40 mg/m² for 5 days), one course every month for 6 months then one course every other month for 12 additional months associated with alpha2a-interferon 4.5 millions units sub-cutaneously three times a week for 18 months.
* Arm B: CHVP + alpha2a-interferon + rituximab. Patients will receive 6 monthly courses of CHVP (cyclophosphamide 600 mg/m², adriamycin 25 mg/m², etoposide 100 mg/m² on day 1 and prednisolone 40 mg/m² for 5 days) associated with 6 infusions of rituximab (375 mg/m2) associated with alpha2a-interferon 4.5 millions units sub-cutaneously three times a week for 18 months.

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed follicular lymphoma with a biopsy performed in the last 3 months
* Patients previously untreated.
* Patients with at least one of the following symptoms requiring initiation of treatment:

  * Bulky disease at study entry according to the Groupe d'Etudes Lymphomes Folliculare (GELF) criteria: nodal or extranodal mass > 7cm in its greater diameter
  * B symptoms
  * Eastern Cooperative Oncology Group (ECOG) performance status (PS) > 1
  * Elevated serum lactate dehydrogenase (LDH) or beta2-microglobulin
  * Involvement of at least 3 nodal sites (each with a diameter greater than 3 cm)
  * Symptomatic splenic enlargement
  * Compressive syndrome
  * Pleural/peritoneal effusion
* Age must be > 18 years and less than 76 years
* Having previously signed a written informed consent form.

Exclusion Criteria:

* Transformation to high-grade lymphoma (secondary to "low-grade" follicular lymphoma).
* Patients without a large tumor burden.
* Patients with prior or concomitant malignancies except non-melanoma skin cancer or adequately treated in situ cervical cancer.
* Poor renal function: Serum creatinine > 150 μmol/L,
* Known HIV infection or active hepatitis B virus (HBV) or hepatitis C virus (HCV) infection.
* Patients with contra-indication to interferon, adriamycin, or rituximab.
* Serious underlying medical conditions, which could impair the ability of the patient to participate in the trial (e.g. ongoing infection, uncontrolled diabetes mellitus, gastric ulcers, active autoimmune disease). Judgment is up to the investigator.
* Known sensitivity or allergy to murine products
* Adult patient under tutelage.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 360
Dates: Start 2000-05; Study Completion 2004-12

PRIMARY OUTCOMES:
Event free survival

SECONDARY OUTCOMES:
Response rate
Overall survival

CONTACTS AND LOCATIONS:
Overall Officials: Gilles A Salles, MD PhD, Principal Investigator — Lymphoma Study Association
Locations (5):
- Groupe d'Etude des Lymphomes de l'adulte, Mont-Godinne, Belgium
- France (4):
  - Hôpital Henri Mondor, Créteil
  - Hôpital Saint Louis, Paris
  - Service d'Hématologie - Centre Hospitalier Lyon-Sud, Pierre-Bénite
  - Centre Henri Becquerel, Rouen

REFERENCES:
- [Background] Solal-Celigny P, Lepage E, Brousse N, Reyes F, Haioun C, Leporrier M, Peuchmaur M, Bosly A, Parlier Y, Brice P, et al. Recombinant interferon alfa-2b combined with a regimen containing doxorubicin in patients with advanced follicular lymphoma. Groupe d'Etude des Lymphomes de l'Adulte. N Engl J Med. 1993 Nov 25;329(22):1608-14. doi: 10.1056/NEJM199311253292203. PMID 8232429
- [Background] McLaughlin P, Grillo-Lopez AJ, Link BK, Levy R, Czuczman MS, Williams ME, Heyman MR, Bence-Bruckler I, White CA, Cabanillas F, Jain V, Ho AD, Lister J, Wey K, Shen D, Dallaire BK. Rituximab chimeric anti-CD20 monoclonal antibody therapy for relapsed indolent lymphoma: half of patients respond to a four-dose treatment program. J Clin Oncol. 1998 Aug;16(8):2825-33. doi: 10.1200/JCO.1998.16.8.2825. PMID 9704735
- [Derived] Salles G, Mounier N, de Guibert S, Morschhauser F, Doyen C, Rossi JF, Haioun C, Brice P, Mahe B, Bouabdallah R, Audhuy B, Ferme C, Dartigeas C, Feugier P, Sebban C, Xerri L, Foussard C. Rituximab combined with chemotherapy and interferon in follicular lymphoma patients: results of the GELA-GOELAMS FL2000 study. Blood. 2008 Dec 15;112(13):4824-31. doi: 10.1182/blood-2008-04-153189. Epub 2008 Sep 17. PMID 18799723
- See also: Official site of the Groupe d'Etudes des Lymphomes de l'Adulte (In french) — http://www.gela.org